CLINICAL TRIAL: NCT00990145
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Multiple-Dose Safety, Tolerability, and Pharmacokinetics Study of EDP-322 in Healthy Adult Volunteers
Brief Title: Multiple Ascending-Dose Study of EDP 322 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Maria T. Madison, Sc.D., Enanta Pharmaceuticals, Inc.
Allocation: Randomized | Masking: Triple
Other Study IDs: EDP-322-07-002
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: MRSA, SSTI

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): EDP-322 v. Placebo
  Interventions: Drug: EDP-322

INTERVENTIONS:
Drug: EDP-322

SUMMARY:
This was a Phase I, single-center, randomized, double-blind, placebo-controlled, ascending multiple dose study to evaluate the safety, tolerability, and pharmacokinetics of orally administered EDP-322 in healthy adult volunteers.

DETAILED DESCRIPTION:
Fifty-two subjects were enrolled into 6 cohorts. Six subjects of each cohort were randomized to received EDP-322 and 2 subjects of each cohort received placebo. Each cohort received the study drug once daily (QD) for 7 days under fed conditions. Multiple oral doses of EDP 322 ranging from 200 to 800 mg were safe and generally well tolerated by the healthy male and female subjects in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females between 18 and 45 years of age
* Females are eligible if documentation exists that they are surgically sterilized
* In good general health [determined by medical history, physical examination, clinical laboratory tests, and without evidence of a clinically significant abnormality, in the opinion of the investigator and medical monitor.
* Subject has a resting 12-lead ECG at screening that shows no clinically significant abnormality and a Bazett-corrected QT interval less than 450 milliseconds.
* BMI between 18-32 kg/m2
* Subject read, understood, and signed the ICF

Exclusion Criteria:

* History of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, CNS, hematologic or metabolic disease, or has an immunologic, emotional, and/or psychiatric disturbance.
* History of gastric surgery, etc.
* Abnormality or clinical lab test results at Screening that is considered clinical significant by the investigator or the medical monitor.
* Gastroenteritis within 1 week before Day 1.
* Acute illness that could pose a threat or harm to the subject or interfere with laboratory test results or interpretation of study data.
* Donated blood within a 4 week period before Day 1.
* Positive for Hep B, C or HIV-1, HIV=2, or positive results at Screening for hepatitis B surface antigen (HBsAG), HCV antibody, or HIV-1 or HIV-2 antibodies
* Medication-related exclusions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The study objective was to determine the safety, tolerability and pharmacokinetics of multiple oral doses of EDP-322 in healthy volunteers. | Subjects received single doses of the study drug administered QD on Days 1 through 7, with follow-up through Day 11, and as needed.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase I Unit, Austin, Texas, United States